CLINICAL TRIAL: NCT02559986
Title: Follow-up of Postpartum Depression After Referral From Pediatric Clinics
Brief Title: Follow up of Mothers Suspected of Postpartum Depression
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nerissa Bauer, Assistant Professor, Indiana University
Other Study IDs: 1111007501
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: telephone interview — telephone interview about their care received during the first year of life and associated events

SUMMARY:
Postpartum depression (PD) is a serious and disabling mental health condition that affects 10-15% of women after childbirth. Low-income minority women are disproportionately affected. Untreated PD can lead to significant negative outcomes for both mother and child. Pediatricians are being asked to routinely screen for PD and while screening rates are improving, little is known about whether mothers actually adhere to pediatrician recommendations to seek additional help after a positive PD screen. The objective of this study is to describe the rate at which mothers seek treatment for suspected PD after a positive screen at the pediatrician office. Additional examination will look at factors that predict whether a mother recalls a recommendation to seek treatment.

DETAILED DESCRIPTION:
The primary outcome of interest is whether mothers suspected of having PD seek treatment after discussion with the pediatrician. In order to evaluate whether discussion with pediatricians leads mothers to seek care, data collection efforts should focus on what information was exchanged, the level of shared decision-making about possible treatment options and whether an agreed upon plan was reached between both parties. The investigators will examine the effectiveness of these discussions by interviewing mothers who were suspected of having PD and referred for treatment. The investigators hypothesize that pediatricians who are able to engage mothers in a shared decision will result in more of those mothers seeking help and getting into appropriate treatment for PD.

The specific research aims of this proposal are to:

Aim 1: Describe the rate at which mothers suspected by pediatricians of having PD seek treatment.

Aim 2: Explore what factors predict whether mothers suspected of PD seek treatment, including maternal sociodemographic characteristics, family centeredness of pediatrician care, and extent of shared decision-making strategy used by the pediatrician.

This will be a cohort study examining the rate at which mothers suspected of having PD seek care and the relationship between shared decision-making and seeking mental health care. Data for both specific aims will be collected by a single telephone interview with mothers suspected of having PD by the pediatrician and referred. For this study, investigators will be focusing recruitment efforts in the four Wishard community health centers (now Eskenazi Health) that use CHICA. In 2007, these four clinics saw 8,528 patients between the ages of 0 and 3 years. These clinics serve a large proportion of families that are underserved, economically disadvantaged and are ethnically and racially diverse.

ELIGIBILITY:
Inclusion Criteria:

-mothers with a positive PD screen who brought their child to seek medical care at participating study clinics, who were present for a majority of the child's visits.

Exclusion Criteria:

-not biological mother, did not bring child to majority of clinic visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mothers whose children received care at one of 4 community general pediatrics clinic with the Child Health Improvement through Computer Automation (CHICA) system who had a positive PD screen and brought the child to the majority of the child's visits to the study clinic
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate at which mothers sought treatment for suspected PD | Within 1 year of index visit
  Defined broadly as a positive response to either called adult care provider (primary care provider, obstetrician, or mental health therapist) for appointment or community resource

SECONDARY OUTCOMES:
Factors associated with help seeking behavior | Within 1 year of index visit
  socio-demographics and other characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Nerissa S Bauer, MD, MPH, Principal Investigator — Indiana University School of Medicine